CLINICAL TRIAL: NCT03303651
Title: Investigation of the Effect of Opioid Titration Guided by Analgesia Indices During General Anesthesia
Brief Title: Monitor-Guided Analgesia During General Anesthesia - Part I
Acronym: MOGADA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20170824
Record Dates: First submitted 2017-08-28; First posted 2017-10-06 (Actual); Last update posted 2018-04-25 (Actual); Status verified 2018-04

CONDITIONS: Pain; Pain, Postoperative; Nociceptive Pain; Opioid Use; Analgesia
Keywords: Analgesia, Monitoring, Opioid, Sufentanil, Sevoflurane
MeSH Terms: conditions — Pain; Pain, Postoperative; Nociceptive Pain; Agnosia | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Participants are assigned to intervention groups by chance
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants are not informed about the group assignement (intervention takes place in general anesthesia). Outcome assessors are persons without knowledge on former treatment in intervention/control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- PPI (Pain Pupillary Index) (Experimental): Opioid administration guided by Pain Pupillary Index (PPI) derived from Videopupillometry performed with the device AlgiScan manufactured by IDMed, Marseille, France. The device measures the degree of pupillary reflex dilation (PRD) following an electric nociceptive stimulation. It automatically increases the intensity of the electric stimulation from 10 to 60 milliampere depending on the degree of PRD and afterwards displays the PPI. The numerical index ranges from 0 to 10. A low PPI score indicates a deep analgesia, a high PPI score indicates an insufficient or light analgesia. A PPI score of 2 or 3 is supposed to represent an optimal level of analgesia according to the manufacturer. 5 µg sufentanil will be administered every 5 minutes if PPI score is calculated more than 3.
  Interventions: Procedure: Opioid administration in intervention groups
- SPI (Surgical Pleth Index) (Experimental): Opioid administration (sufentanil) guided by by Surgical Pleth Index (SPI) derived from photoplethysmography performed by the device CARESCAPE B650 Patient Monitor from the manufacturer GE (General Electrics) Healthcare, Helsinki, Finland. Included in the monitoring system is a software that continuously calculates the SPI from normalized heart rate and pulse wave amplitude derived from finger plethysmography. The numerical index ranges between 0 (low sympathetic tone) and 100 (high sympathetic tone). A SPI score between 20 and 50 has been proposed as the target range to guide analgesics (15 - 17). 5 µg Sufentanil will be administered every 5 minutes if SPI score is calculated more than 50.
  Interventions: Procedure: Opioid administration in intervention groups
- NOL (Nociception Level) (Experimental): Opioid administration (sufentanil) guided by Nociception Level (NOL) derived from finger photoplethysmography performed with the analgesia monitoring device PMD200 manufactured by Medasense, Ramat Gan, Israel. The device continuously calculates the NOL with a multi-parametric approach from pulse rate, pulse rate variability, pulse wave amplitude, skin conductance level, skin conductance fluctuations, skin temperature and finger motion. The composite algorithm of the device analyses the data and the numerical index NOL is presented on a scale from 0 (no pain) to 100 (extreme pain) (18). A NOL score between 10 and 25 has been proposed as the target range to guide analgesics. 5 µg Sufentanil will be administered every 5 minutes if NOL score is calculated more than 25.
  Interventions: Procedure: Opioid administration in intervention groups
- Control (Active Comparator): Opioid administration (sufentanil) guided according to standard clinical practice of the attending anesthesiologist based upon changes of heart rate, blood pressure, lacrimation and sweating of the patient.
  Interventions: Procedure: Opioid administration in control group

INTERVENTIONS:
Procedure: Opioid administration in intervention groups — Elective surgery in radical open abdominal prostatectomy. Opioid titration is guided by analgesia indices during general anesthesia in the experimental arms.
  Arms: NOL (Nociception Level); PPI (Pain Pupillary Index); SPI (Surgical Pleth Index)
Procedure: Opioid administration in control group — Elective surgery in radical open abdominal prostatectomy. Opioid titration is guided by clinical signs in the control group.
  Arms: Control

SUMMARY:
This prospective randomized clinical trial evaluates the effects of a monitor-guided opioid analgesia during general anesthesia. To date no standard-monitoring device exists to specifically reflect the analgesic component of general anesthesia. Quality and safety of general anesthesia are of major clinical importance and should be improved by limiting the opioid analgesic's dosage to the minimum amount needed. The study compares the effects of monitoring nociception during general anesthesia with different innovative techniques in comparison to routine clinical practice.

DETAILED DESCRIPTION:
This prospective randomized clinical study aims to investigate the effects of a monitor-guided opioid analgesia during general anesthesia by different monitoring systems in comparison to routine clinical practice. Many surgical procedures require general anesthesia. The main components of general anesthesia are hypnosis and analgesia, and anesthesiologists usually combine a hypnotic drug with an opioid analgesic.

Until today, however, there is no standard-monitoring of nociception to specifically reflect the analgesic component of general anesthesia. In clinical practice the opioid dosage is chosen by clinical judgment of the attending anesthesiologist based upon changes of heart rate, blood pressure, pupil size, lacrimation and sweating of the patient.

On the one hand, underdosage of opioids can cause nociception leading to an increased sympathetic tone, increase of plasma levels of stress hormones, nociceptive movements as well as increase postoperative pain. On the other hand, overdosage of opioids can lead to drug side effects such as nausea and vomiting, hemodynamic instability, an increase in recovery times, immunosuppression and an increase in postoperative pain by opioid-induced-hyperalgesia. Quality and safety of general anesthesia are of major clinical importance and can be improved by limiting the administration of opioid analgesics to the optimal individual dose needed. In the last years, different analgesia monitoring devices have been developed for monitoring nociception. The present study evaluates the effects of the administration of opioids during general anesthesia guided by three different monitoring systems in comparison to routine clinical practice. After institutional approval by the Ethics committee of the Medical Board of the City of Hamburg, Germany and obtaining patients' written informed consent the investigators randomize elective patients with major abdominal surgery for open radical prostatectomy into one of four treatment groups.

ELIGIBILITY:
Inclusion Criteria:

* Radical open abdominal prostatectomy scheduled in the operation theater where the study is conducted
* > 18 years

Exclusion Criteria:

* Chronic pain therapy, e.g. out-of-hospital opioid therapy
* Beta blocker and digitalis therapy
* Eye disease with affection of pupil reactivity
* Pacemaker therapy
* Higher degrees of cardiac arrhythmias, e.g. atrial fibrillation
* Pre-operative medication with steroids

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2017-10-16 (Actual); Primary Completion 2017-12-05 (Actual); Study Completion 2018-01-26 (Actual)

PRIMARY OUTCOMES:
Intraoperative opioid consumption | 1 day
  Compares the amount of intraoperative opioid administration (sufentanil) per minute of general anesthesia and per kg bodyweight between groups.

SECONDARY OUTCOMES:
Time to extubation | 1 day
  Postoperative recovery time: Time interval between end of operation and tracheal extubation of the patient.
Time to fit-for-discharge | 1 day
  Postoperative recovery time: Time interval between postoperative tracheal extubation and the patient reaching fit-for-discharge criteria from the PACU to the ward.
Postoperative pain level | 1 day
  Postoperative pain level measured with the highest score in numeric pain rating scale (NRS).
Postoperative opioid administration | 1 day
  Amount of postoperative opioid administration (piritramid) in the postanesthesia care unit (PACU). Piritramid is given if NRS score is > 3.
Patient satisfaction | 2-21 days
  Patient satisfaction with the general anesthesia and pain management evaluated by a numeric rating scale.
Release of stress hormones | 1 day
  Amount of perioperative plasma level of cortisol and ACTH.

CONTACTS AND LOCATIONS:
Overall Officials: Rainer Nitzschke, MD, Principal Investigator — Department of Anesthesiology; Center of Anesthesiology and Intensive Care Medicine, Hamburg Eppendorf University Medical Center; Sandra Funcke, MD, Principal Investigator — Department of Anesthesiology; Center of Anesthesiology and Intensive Care Medicine, Hamburg Eppendorf University Medical Center
Locations (1):
- Department of Anesthesiology; Center of Anesthesiology and Intensive Care Medicine, Hamburg Eppendorf University Medical Center, Hamburg, Germany

IPD SHARING:
Plan to Share IPD: No
All data will be anonymized before publication.